CLINICAL TRIAL: NCT04326725
Title: Proflaxis for Healthcare Professionals Using Hydroxychloroquine Plus Vitamin Combining Vitamins C, D and Zinc During COVID-19 Pandemia: An Observational Study
Brief Title: Proflaxis Using Hydroxychloroquine Plus Vitamins-Zinc During COVID-19 Pandemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Mehmet Mahir Ozmen, Professor of Surgery, Department of Surgery, Istinye University
Other Study IDs: 2020-2/1
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Pneumonitis; Coronavirus Infection
Keywords: Hydroxychloroquine; coronavirus; prophylaxis; healthcare professional; outbreak
MeSH Terms: conditions — Pneumonia; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hydroxychloroquine: Subjects with prophylaxis
  Interventions: Drug: Plaquenil 200Mg Tablet

INTERVENTIONS:
Drug: Plaquenil 200Mg Tablet — health workers under risk who took this medications
  Other Names: Redoxan

SUMMARY:
Healthcare professionals mainly doctors, nurses and their first degree relatives (spouse, father, mother, sister, brother, child) who have been started hydroxychloroquine(plaquenil) 200mg single dose repeated every three weeks plus vitaminC including zinc once a day were included in the study. Study has conducted on 20th of march. Main purpose of the study was to cover participants those who are facing or treating COVID19 infected patients in Ankara.

DETAILED DESCRIPTION:
Healthcare professionals mainly doctors, nurses and their first degree relatives (spouse, father, mother, sister, brother, child) who have been started hydroxychloroquine(plaquenil) 200mg single dose repeated every three weeks plus vitaminC including zinc once a day were included in the study. Study has conducted on 20th of march. Main purpose of the study was to cover participants those who are facing or treating COVID19 infected patients.PArticipants, age, sex, BMI, smoking history, comorbid disease were also registered.

ELIGIBILITY:
Inclusion Criteria:

1. person who are working as health professional with contact to known COVID positive case
2. Their first degree relatives (child, spouse or parents)
3. must be able to swallow tablets

Exclusion Criteria:

1. Already using plaquenil for other reasons (RA etc)
2. person with the diagnosis of COVID infection
3. Person with the condition may cause complications with this medication (severe CVD, av block, already has ophtalmological complications, organ failure of any degree etc).
4. Documented allergic history to chloroquine;
5. Documented history of hematological system diseases;
6. Documented history of chronic liver and kidney diseases;
7. Documented history of cardiac arrhythmia or chronic heart diseases;
8. Documented history of retina or hearing dysfunction;
9. Documented history of mental illnesses; 10. Use of digitalis due to the previous disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mainly doctors, nurses, health workers in the hospital whereby they have close contacts with possile COVID-19 infected patients were included. Their first degree relatives(spouse, child, parents)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Protection against COVID-19 | 4 months
  persons who took this medication should not have an infection

CONTACTS AND LOCATIONS:
Overall Officials: Mahir M Ozmen, Professor, Principal Investigator — Istinye University
Locations (1):
- Istinye University Medical School, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Dong L, Hu S, Gao J. Discovering drugs to treat coronavirus disease 2019 (COVID-19). Drug Discov Ther. 2020;14(1):58-60. doi: 10.5582/ddt.2020.01012. PMID 32147628
- [Background] Kruse RL. Therapeutic strategies in an outbreak scenario to treat the novel coronavirus originating in Wuhan, China. F1000Res. 2020 Jan 31;9:72. doi: 10.12688/f1000research.22211.2. eCollection 2020. PMID 32117569
- [Background] Song P, Karako T. COVID-19: Real-time dissemination of scientific information to fight a public health emergency of international concern. Biosci Trends. 2020 Mar 16;14(1):1-2. doi: 10.5582/bst.2020.01056. Epub 2020 Feb 25. PMID 32092748
- [Background] Lake MA. What we know so far: COVID-19 current clinical knowledge and research. Clin Med (Lond). 2020 Mar;20(2):124-127. doi: 10.7861/clinmed.2019-coron. Epub 2020 Mar 5. PMID 32139372
- [Background] Cunningham AC, Goh HP, Koh D. Treatment of COVID-19: old tricks for new challenges. Crit Care. 2020 Mar 16;24(1):91. doi: 10.1186/s13054-020-2818-6. No abstract available. PMID 32178711
- [Background] Plantone D, Koudriavtseva T. Current and Future Use of Chloroquine and Hydroxychloroquine in Infectious, Immune, Neoplastic, and Neurological Diseases: A Mini-Review. Clin Drug Investig. 2018 Aug;38(8):653-671. doi: 10.1007/s40261-018-0656-y. PMID 29737455